CLINICAL TRIAL: NCT06689969
Title: Evaluation of the Effect of Osseodensification on the Peri-implant Condition
Brief Title: Effect of Osseodensification on the Peri-implant Condition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asem Mohammed Kamel Ali, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Osseodensification in implant
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Implant Therapy
Keywords: Osseodensification

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with narrow ridge received small diameter implant in conventional method. (Active Comparator)
  Interventions: Procedure: conventional implant placement method
- patients with narrow ridge received implant by OD technique using densah bur. (Active Comparator)
  Interventions: Procedure: Osseodensification to implant placement using densah bur kit

INTERVENTIONS:
Procedure: conventional implant placement method — Site marking was the first step in preparing the place for implantation. Subsequently, using a high speed surgical handpiece and a surgical motor, a pilot drill was revolved at 1200 RPM in a clockwise rotation to the desired depth, creating a 1.5 mm first pilot osteotomy. An X-ray was obtained using paralleling pins to validate the angle between the surrounding teeth and the implants. Eventually the implant's precise placement was established. To prepare the osteotomy site to the desired diameter, drills are used sequentially at 1200 RPM in a clockwise motion. Gradually bigger drill diameters were used for incremental drilling. Based on the diameter of the desired implant, bur sizes were utilized in ascending order
  Arms: patients with narrow ridge received small diameter implant in conventional method.
Procedure: Osseodensification to implant placement using densah bur kit — Beginning with site marking, the area was prepared for implantation. A high speed surgical handpiece and a surgical motor (surgic pro® NSK, Japan) were then used to construct a 1.5 mm initial pilot osteotomy using a pilot drill spun at 1200 RPM in a clockwise rotation to the desired depth. In order to verify the angle between the surrounding teeth and the implants, paralleling pins were used to capture an X-ray.
  After it was determined that the implant was in the proper location, OD was used to extend the osteotomy using a Densah® Bur VT1525 2.0-mm (VersahTM, LLC, USA) in non-cutting anticlockwise rotation at 1200 RPM (Densifying Mode). The osteotomy was expanded to the desired diameter by repeatedly using a DensahTM Bur operating in a non-cutting anticlockwise (CCW) direction at 1200 RPM (Densifying Mode). Gradually increasing drill diameters were used for incremental drilling. Based on the diameter of the desired implant, bur sizes (diameters) were utilised in ascending order
  Arms: patients with narrow ridge received implant by OD technique using densah bur.

SUMMARY:
The goal of this clinical trial is to evaluate the effects of osseodensification vs. traditional implant site preparation clinically , radiographically, bio-chemically. in patients of both sexes, ages 25 to 45, who had bilaterally missed maxillary teeth. The main questions it aims to answer are :which technique was the better results give at implant placement? Researchers will compare Osseodensification maneuver in implant placement to see if implant stability increased also peri-implant tissue accurately formed or the same in traditional implant site preparation. Participants will receiving dental implants in narrow maxillary posterior ridge via small diameter implant in conventional method in first entity while in second entity implant by osseodensification technique using densah bur.

ELIGIBILITY:
Inclusion Criteria:

* All patients were free from any systemic diseases
* Individuals above age of 18 who have thin ridges and missing bilateral maxillary posterior teeth

Exclusion Criteria:

* Severe skeletal discrepancy.
* Para functional habits.
* Patients who had already received or lost implants in the potential implantation site.
* Smoker patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Implant primary stability | A single time point (once immediately after implant placement)
  Osstell® Mentor magnetic resonance instrument used to measure primary stability
Bone density | From enrollment to the end of treatment at 24 weeks" (at the beginning, one, three-, and six-months following implant insertion)
  Measuring of bone density (BD) through using the image J analysis software application
Assessment of interleukin -6 | From enrollment to the end of treatment at 24 weeks" (at the beginning, one, three-, and six-months following implant insertion)
Assessment of Vascular endothelial growth factor | [Time Frame: From enrollment to the end of treatment at 24 weeks" (at the beginning, one, three-, and six-months following implant insertion)]

SECONDARY OUTCOMES:
Peri-implant probing depth | From enrollment to the end of treatment at 24 weeks" (at the beginning, three-, and six-months following implant insertion)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dental medicine, Al-Azhar University (Assiut branch), Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strietzel FP, Nowak M, Kuchler I, Friedmann A. Peri-implant alveolar bone loss with respect to bone quality after use of the osteotome technique: results of a retrospective study. Clin Oral Implants Res. 2002 Oct;13(5):508-13. doi: 10.1034/j.1600-0501.2002.130510.x. PMID 12453128
- [Background] Johnson RB, Serio FG, Dai X. Vascular endothelial growth factors and progression of periodontal diseases. J Periodontol. 1999 Aug;70(8):848-52. doi: 10.1902/jop.1999.70.8.848. PMID 10476891
- [Background] Trisi P, Berardini M, Falco A, Podaliri Vulpiani M. New Osseodensification Implant Site Preparation Method to Increase Bone Density in Low-Density Bone: In Vivo Evaluation in Sheep. Implant Dent. 2016 Feb;25(1):24-31. doi: 10.1097/ID.0000000000000358. PMID 26584202